CLINICAL TRIAL: NCT06754332
Title: The Research on the Role of Human Chorionic Gonadotropin (HCG) Activation in Vivo on the Dormant Follicles in Patients With Premature Ovarian Insufficiency (POI).
Brief Title: The Study of Human Chorionic Gonadotropin (HCG) Activating the Dormant Follicles .
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KY-2024-242
Record Dates: First submitted 2024-12-24; First posted 2024-12-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Premature Ovarian Insufficiency
Keywords: POI; HCG; dormant follicles
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Expectant treatment (No Intervention): The POl patients undergo transvaginal ultrasound to observe follicular growth every 1-2 weeks, with a monitoring period of 3 months.
- In vitro fertilization - Embryo transfer (Other): Embryo vitrification and freezing were performed after fertilization of oocytes.
  Interventions: Drug: human chorionic gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin — The POI patients receive a single intramuscular injection of 10,000 units of human chorionic gonadotropin.
  Other Names: HCG
  Arms: In vitro fertilization - Embryo transfer

SUMMARY:
This project aims to activate dormant follicles in patients with premature ovarian insufficiency by injecting human chorionic gonadotropin (hCG) to explore the feasibility of a treatment plan that stimulates the growth of dormant follicles, not visible to the naked eye, to antral follicles visible under ultrasound, without visible follicle growth. The project also seeks to enable patients to conceive offspring carrying their own genetic material through in vitro fertilization (IVF) technology.

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Females under 40 years of age with amenorrhea or oligomenorrhea for at least four months, and elevated follicle-stimulating hormone (FSH) levels > 25 IU/l on two separate occasions (with a 4-week interval);
2. Ultrasound (B-mode) indicating no antral follicle development in both ovaries for at least 3 months prior to study participation;
3. Those who agree to participate in this study and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Individuals over 40 years of age, or under 40 years of age with regular menstruation, normal ovulation, amenorrhea or oligomenorrhea for less than 4 months, and elevated follicle-stimulating hormone (FSH) levels < 25 IU/l on two or more separate occasions (with a 4-week interval);
2. Those with contraindications to the use of injectable human chorionic gonadotropin (HCG);
3. Those with asthma, epilepsy, heart disease, migraines, renal impairment, hypertension, or other diseases;
4. Patients deemed by the researcher as otherwise unsuitable for participation in this study.

Withdrawal criteria:

1. Subjects who cannot follow up as scheduled or have poor compliance with the experimental treatment;
2. Significant safety events occur, and the investigator deems it necessary for the subject to withdraw.Study Method: A total of 60 patients with premature ovarian insufficiency who are planned to undergo in vitro fertilization (IVF) treatment at our hospital were included. Patients were divided into two groups based on their consent to receive HCG injection: the control group (those who did not agree to HCG injection) and the HCG group (those who agreed to HCG injection).

The HCG group received a single intramuscular injection of 10,000 units of HCG. One to two weeks after the injection, transvaginal ultrasound was performed to observe follicular growth, with a monitoring period of 3 months (based on the fact that it takes humans 85 days to develop from a secondary follicle to a mature follicle). If no follicular growth was observed within 3 months, the observation was abandoned. If follicular growth was observed, gonadotropins were used or not used based on follicular development to promote growth or antagonists were used to prevent premature follicular release. When the follicle reached ≥18mm and estradiol reached ≥150pg/ml, recombinant human chorionic gonadotropin (rhCG) 250ug and triptorelin 0.1mg were co-administered to trigger ovulation. Oocyte retrieval was performed 36 hours after triggering. If embryos were obtained, they were cryopreserved for later frozen-thawed embryo transfer (FET) assistance in conception.

The control group underwent transvaginal ultrasound to observe follicular growth every 1-2 weeks, with a monitoring period of 3 months. If no follicular growth was observed within 3 months, the observation was abandoned. If follicular growth was observed, gonadotropins were used or not used based on follicular development to promote growth or antagonists were used to prevent premature follicular release. When the follicle reached ≥18mm and estradiol reached ≥150pg/ml, rhCG 250ug and triptorelin 0.1mg were co-administered to trigger ovulation. Oocyte retrieval was performed 36 hours after triggering. If embryos were obtained, they were cryopreserved for later FET assistance in conception.

Follow-up Plan: ① Within 3 months after HCG administration, patients return to the center every 1-2 weeks for ultrasound and hormone testing, and return to the hospital promptly if any discomfort occurs during this period. ② After embryo transfer and pregnancy, follow-up on the outcome of childbirth, and follow-up on the offspring until one year after birth.

ELIGIBILITY:
Inclusion Criteria:

1. Females under 40 years of age with amenorrhea or oligomenorrhea for at least four months, and elevated follicle-stimulating hormone (FSH) levels > 25 IU/l on two separate occasions (with a 4-week interval);
2. Ultrasound (B-mode) indicating no antral follicle development in both ovaries for at least 3 months prior to study participation;
3. Those who agree to participate in this study and voluntarily sign the informed consent form.

Exclusion Criteria:

1. Individuals over 40 years of age, or under 40 years of age with regular menstruation, normal ovulation, amenorrhea or oligomenorrhea for less than 4 months, and elevated follicle-stimulating hormone (FSH) levels < 25 IU/l on two or more separate occasions (with a 4-week interval);
2. Those with contraindications to the use of injectable human chorionic gonadotropin (HCG);
3. Those with asthma, epilepsy, heart disease, migraines, renal impairment, hypertension, or other diseases;
4. Patients deemed by the researcher as otherwise unsuitable for participation in this study."

Ages: 20 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
focilles | Interval of 1-2 weeks after HCG injection
  Bilateral ovarian follicles were monitored by ultrasound

SECONDARY OUTCOMES:
sex hormone | Interval of 1-2 weeks after HCG injection
  chemiluminescence method
Oocyte | After the egg retrieval operation, the eggs are picked up and observed
  Stereo microscope
Embryo | 3-5 days after In vitro fertilization
  Stereo microscope
Pregnancy outcome | One month after embryo transfer
  Ultrasonic
The health of the offspring | One year after birth
  Telephone follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Chen, Master, Principal Investigator — The Fourth Affiliated Hospital Zhejiang University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Xiao Y, Peng X, Peng Y, Zhang C, Liu W, Yang W, Dou X, Jiang Y, Wang Y, Yang S, Xiang W, Wu T, Li J. Macrophage-derived extracellular vesicles regulate follicular activation and improve ovarian function in old mice by modulating local environment. Clin Transl Med. 2022 Oct;12(10):e1071. doi: 10.1002/ctm2.1071. PMID 36229897
- [Result] Cha KY, Chian RC. Maturation in vitro of immature human oocytes for clinical use. Hum Reprod Update. 1998 Mar-Apr;4(2):103-20. doi: 10.1093/humupd/4.2.103. PMID 9683349
- [Result] Chian RC, Li JH, Lim JH, Yoshida H. IVM of human immature oocytes for infertility treatment and fertility preservation. Reprod Med Biol. 2023 Jul 11;22(1):e12524. doi: 10.1002/rmb2.12524. eCollection 2023 Jan-Dec. PMID 37441160